CLINICAL TRIAL: NCT03833128
Title: An Open Label Study to Determine the Safety and Tolerability of 12 Weeks Treatment With Oral REN001 in Subjects With Fatty Acid Oxidation Disorders (FAOD)
Brief Title: A Phase 1b Study of the Safety of REN001 in Patients With Fatty Acid Oxidation Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reneo Pharma Ltd (Industry)
Responsible Party: Sponsor
Organization: OnKure, Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: REN001-102
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Fatty Acid Oxidation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 - Part A (Experimental): REN001 Low Dose oral once daily x 12 weeks
  Interventions: Drug: Low Dose REN001
- Group 2 - Part A (Experimental): REN001 High Dose oral once daily x 12 weeks
  Interventions: Drug: High Dose REN001
- Group 3 - Part B (Experimental): REN001 High Dose oral once daily x 12 weeks
  Interventions: Drug: High Dose REN001

INTERVENTIONS:
Drug: Low Dose REN001 — Oral
  Arms: Group 1 - Part A
Drug: High Dose REN001 — Oral
  Arms: Group 2 - Part A; Group 3 - Part B

SUMMARY:
The purpose of this Phase 1b study is to assess REN001 safety in subjects with fatty acid oxidation disorders.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, multiple-dose study of the safety and tolerability of 2 dose levels of REN001 in subjects with fatty acid oxidation disorders (FAODs) with confirmed mutations in the Carnitine palmitoyltransferase II deficiency (CPT2), Very long-chain Acyl-CoA dehydrogenase deficiency (VLCAD), Long-chain 3-hydroxyacyl-CoA dehydrogenase deficiency (LCHAD) or Trifunctional Protein Deficiency (TFP). All subjects will provide written consent prior to commencing any study related activities or assessments. Potential subjects will be screened for study participation up to 8 weeks prior to the start of dosing.The study is divided into two parts, Part A and Part B. Part A has finished enrollment and further eligible patients will participate in Part B only.

ELIGIBILITY:
Inclusion Criteria:

Subjects must give written, signed and dated informed consent

Confirmed diagnosis of FAOD

A diagnostic acylcarnitine profile, in blood or cultured fibroblasts

A stable treatment regimen for at least 30 days prior to enrollment

Exclusion Criteria:

Unstable or poorly controlled disease

Treatment with an investigational drug within 1 month or within 5 half-lives, whichever is longer

Have been hospitalized within 3 months prior to screening for any major medical event

Pregnant or nursing females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Continous to Week 12
  Number of participants with Adverse Events (AEs) as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Vockley, M.D., Ph.D., Principal Investigator — University of Pittsburgh Medical Center
Locations (7):
- United States (5):
  - Children's Hospital Colorado, Aurora, Colorado
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Division of Medical Genetics, University Utah, Salt Lake City, Utah
- Neurology department, Raymond-Poincaré Teaching Hospital, Nord/Est/Ile de France Neuromuscular Reference Center, Garches, France
- Servicio de Neurología - Unidad de Neuromuscular Centro de Referencia Nacional de Enfermedades Neuromusculares raras Instituto de Investigación i+12, Madrid, Spain